CLINICAL TRIAL: NCT00641264
Title: Laryngopharyngeal Reflux Health Related Quality of Life (LPR-HRQL) Questionnaire Development and Psychometric Testing in Patients Receiving Omeprazole 20 mg Bid as Treatment for Laryngopharyngeal Reflux.
Brief Title: Quality of Life Validation in Laryngitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, Astra Zeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 294
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Laryngopharyngeal Reflux (LPR)
Keywords: Laryngopharyngeal reflux (LPR); Omeprazole; Losec; Quality of Life; Laryngitis
MeSH Terms: conditions — Laryngopharyngeal Reflux; Laryngitis | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Omeprazole
  Other Names: Losec
Behavioral: Quality of Life questionnaire

SUMMARY:
The primary purpose of this study was to establish the psychometric properties of a new disease specific Quality of Life questionnaire, the LPR-HRQL. The specific properties of the questionnaire that were evaluated were: validity, reliability, and responsiveness to change (as a measure of treatment effect).

ELIGIBILITY:
Inclusion Criteria:

* New Laryngopharyngeal reflux diagnosis less than 1 month or relapsed patients not under current treatment

Exclusion Criteria:

* Unable to comply with study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2001-05; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
LPR-HRQL questionnaire, which measured symptom distress and the effects of LPR on voice, cough, throat clearing, swallow , and overall impact of acid reflux | 2 monthly

SECONDARY OUTCOMES:
Safety assessments via adverse event recording and physical examinations | 2 monthly

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca